CLINICAL TRIAL: NCT01053754
Title: Optimization of the Evaluation of the Adrenal Function After Discontinuation of a Prolonged Therapy With Corticosteroids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/23; 2009-015730-30
Record Dates: First submitted 2010-01-18; First posted 2010-01-21 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Adrenocortical Insufficiency
Keywords: adrenocortical insufficiency; prolonged corticotherapy
MeSH Terms: conditions — Addison Disease

INTERVENTIONS:
Biological: "long" synacthen stimulation test — IM injection of 1 mg of delate synacthen which can be realized in ambulatory conditions

SUMMARY:
The study (forward-looking and opened) will concern 70 subjects having had a systemic prolonged treatment with corticosteroids for intestinal chronic inflammatory disease, recruited in the services of gastroenterology and endocrinology of the North Hospital of Marseille (France). The primary objective of the study is to estimate a new test, the "long" synacthen stimulation test, using an IM injection of 1 mg of delate synacthen, with regard to the definitive standard. Indeed, this long test could be realized in ambulatory conditions, and turn out more contributory than the definitive standard to estimate the capacities of answer of the adrenal glands in front of a prolonged stress, as it is the case during a surgical procedure for example.

The secondary objectives are: 1) to determine the relation between the value of basal cortisol and the peak of stimulation of cortisol during short and long tests. This could allow to clarify better the conditions in which it is absolutely necessary to realize a dynamic test, 2) to determine the relation between cortisol assay in the plasma and in the saliva. The sample of saliva is simple and non-invasive, and presents the advantage to be able to be realized in ambulatory conditions and by the patient himself.

The cortisonic withdrawal syndrome is another complication which can arise when a prolonged corticosteroid therapy is discontinued. Clinically, it looks like a chronic adrenocortical insufficiency, but with normal ranges of plasma cortisol. It is probably in touch with a physical dependence to the taking of above physiological doses of GC over a long period. Its physiopathology remains badly known, but could bring in a deficit of secretion of DHEA-S (dehydro-epiandrosterone sulphate), another hormone secreted by the adrenal glands. One of the secondary objectives of the study will consist in informing the variations of DHEA-S after a prolonged corticotherapy, in the basal state and after stimulation by the long synacthen stimulation test.

DETAILED DESCRIPTION:
Synthetic glucocorticoids (GC) are used in the treatment of numerous inflammatory or auto-immune diseases, in particular the intestinal chronic inflammatory diseases (Crohn's disease, chronic ulcerative colitis). In case of discontinuation of a prolonged (superior to 3-4 weeks) and systemic treatment, deleterious side effects are frequent, with in particular a risk of adrenocortical insufficiency and withdrawal cortisonic syndrome. Our protocol of medical research concerns these two complications, and aims at optimizing the evaluation of the adrenal function.

The adrenocortical insufficiency after prolonged corticotherapy is the most frequent cause of secondary adrenocortical insufficiency. It is due to the braking of the hypothalamo-pituitary-adrenal (HPA) axis which controls the endogenous secretion of cortisol. It is mostly transient, but can last several months, and exposes to a risk of acute decompensation. An adapted coverage with replacement doses of hydrocortisone (natural GC) is thus necessary during the treatment discontinuation, together with regular hormonal revaluations to track down the recovery of the adrenal function. These evaluations are based on biological measurements, because of the absence of specific clinical symptoms. At first, basal plasma cortisol at 08:00 am (physiological peak of the hormone) is assayed. A value lower than 8 µg / dl (220 nmol / l) allows to do the positive diagnosis of adrenal insufficiency and a value superior to 20 µg / dl (550 nmol / l) to exclude it. Between these 2 values, a doubt remains on the capacities of the adrenal glands to secrete enough cortisol in case of stress, and the realization of a dynamic test of stimulation is then necessary. The standard test used in common practice is the "short" synacthene stimulation test (fragment 1-24 of the ACTH, the hormone secreted by the pituitary gland and stimulating the secretion of cortisol) using an IV injection of 250 µg of immediate synacthen. The study (forward-looking and opened) will concern 70 subjects having had a systemic prolonged treatment with corticosteroids for intestinal chronic inflammatory disease, recruited in the services of gastroenterology and endocrinology of the North Hospital of Marseille (France). The primary objective of the study is to estimate a new test, the "long" synacthen stimulation test, using an IM injection of 1 mg of delate synacthen, with regard to the definitive standard. Indeed, this long test could be realized in ambulatory conditions, and turn out more contributory than the definitive standard to estimate the capacities of answer of the adrenal glands in front of a prolonged stress, as it is the case during a surgical procedure for example.

The secondary objectives are: 1) to determine the relation between the value of basal cortisol and the peak of stimulation of cortisol during short and long tests. This could allow to clarify better the conditions in which it is absolutely necessary to realize a dynamic test, 2) to determine the relation between cortisol assay in the plasma (classically used) and in the saliva ( which is validated for the evaluation of the other adrenal pathology as the Cushing's syndrome, but not still in the adrenocortical insufficiency after prolonged corticotherapy). The sample of saliva is simple and non-invasive, and presents the advantage to be able to be realized in ambulatory conditions and by the patient himself.

The cortisonic withdrawal syndrome is another complication which can arise when a prolonged corticosteroid therapy is discontinued. Clinically, it looks like a chronic adrenocortical insufficiency, but with normal ranges of plasma cortisol. It is probably in touch with a physical dependence to the taking of above physiological doses of GC over a long period. Its physiopathology remains badly known, but could bring in a deficit of secretion of DHEA-S (dehydro-epiandrosterone sulphate), another hormone secreted by the adrenal glands. One of the secondary objectives of the study will consist in informing the variations of DHEA-S after a prolonged corticotherapy, in the basal state and after stimulation by the long synacthen stimulation test.

ELIGIBILITY:
Inclusion Criteria:

* Intestinal chronic inflammatory diseases (Crohn's disease, chronic ulcerative colitis)
* Systemic prolonged treatment with corticosteroids during 2 months at least
* Discontinuation of the treatment with corticosteroids for 6 weeks
* Basal plasma cortisol between 8 and 20 µg / dl (220 to 550 nmol / l).

Exclusion Criteria:

* Systemic prolonged treatment with corticosteroids because of an other disease than a intestinal chronic inflammatory disease
* Pregnancy, breast feeding
* Hypersensibility to synacthene
* Basal plasma cortisol lower than 8 µg / dl (220 nmol / l) or superior to 20 µg / dl (550 nmol / l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To estimate a new test, the "long" synacthen stimulation test, using an IM injection of 1 mg of delate synacthen, with regard to the definitive standard. | 2 years

SECONDARY OUTCOMES:
To determine the relation between the value of basal cortisol and the peak of stimulation of cortisol during short and long tests - to determine the relation between cortisol assay in the plasma and in the saliva | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine BOULLU, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France, France